CLINICAL TRIAL: NCT03089970
Title: Using Breath Metabolites to Determine Specific Virus Infection in Asthmatic Patients
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 637013; 1K23HL127185-01A1 (NIH)
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Upper Respiratory Tract Infections, Asthma, Exhaled Breath
MeSH Terms: conditions — Respiratory Tract Infections; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy asthma: Asthmatic patients not with an exacerbation, i.e., stable asthmatics
  Interventions: Diagnostic Test: Exhaled breath condensate collection
- Rhinovirus-infected asthmatics: Asthmatics with an exacerbation and associated rhinovirus infection
  Interventions: Diagnostic Test: Exhaled breath condensate collection
- Influenza A-infected asthmatics: Asthmatics with an exacerbation and associated influenza A infection
  Interventions: Diagnostic Test: Exhaled breath condensate collection

INTERVENTIONS:
Diagnostic Test: Exhaled breath condensate collection — Breath from humans is cooled, condensed, and collected

SUMMARY:
Respiratory virus infections cause a majority of asthma exacerbations in the fall to spring months. Current diagnostic platforms for respiratory viruses have limitations including cost, availability, and invasiveness. The use of noninvasive breath collection to analyze breath metabolites may be used to differentiate virus-infected asthmatics from other causes of acute asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Asthma, Age ≥12, Symptoms/signs of an early asthma exacerbation, Ability to provide exhaled breath condensate (EBC) x15 min, Body mass index (BMI) ≥18

Exclusion Criteria:

* Chronic lung diseases other than asthma (e.g., chronic obstructive pulmonary disease [COPD], lung cancer, fibrotic lung disease, etc.), Smoking in the past 7 days, Eating or non-clear liquids <4 hrs prior to EBC collection, Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with asthma with or without an acute exacerbation will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Breath metabolite differences between groups | 36 months
  Metabolites from breath will be identified and quantified using gas chromatography-mass spectrometry; these will be compared between groups. Specific breath metabolites include isoprostane, linear and branched alkanes (C6-C9), alcohols, and thiol-containing moieties. However, we will also measure metabolites in an un-targeted manner.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schivo, MD, MAS, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Ceneter, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No